CLINICAL TRIAL: NCT06487689
Title: Oral Manifestations in Chronic Kidney Disease: Clinical Trial
Brief Title: Oral Manifestations in Chronic Kidney Disease.
Status: Completed | Type: Observational
Sponsor: José López Lopez (Other)
Responsible Party: Sponsor-Investigator, José López Lopez, doctor, University of Barcelona
Organization: University of Barcelona (Other)
Other Study IDs: Renal-Oral
Record Dates: First submitted 2024-06-12; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Diseases; Hemodyalysis; Pre-dyalisis; Peritoneal Dyalisis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hemodyalisis
- Peritoneal dyalisis
- Pre-dyalisis

SUMMARY:
The goal of this observational study is to investigate oral manifestations in patients with Chronic Kidney Disease (CKD) for early detection, that alterations play an important point for dental guide during the progression and type of treatment of CKD .

An oral exam was performed for detection oral manifestations, age, smoking, alcoholic and oral hygiene habits were collected.

The study has 3 groups under study: hemodialysis (HD), peritoneal dialysis (PD) and pre-dialysis (P-D)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years;
* No change of medication in the last 3 months;
* History of CKD comported by data laboratory (GRF<60 ml/min/1.73m²).

Exclusion Criteria:

* Age ≤ 18 years and ≥ 80 years;
* Patients undergoing orthodontic therapy;
* Patients taking drugs;
* Patients changes the medication or introduced a new medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population with Chronic Kidney Disease, in pre-dialysis, hemodialysis, peritoneal dialysis
Sampling Method: Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Periodontal status | 2 years
  periodontrogram (probe CP12)

SECONDARY OUTCOMES:
Sex | 2 years
  qualitative variable: Male/Female
Age | 2 years
  nominal variable: years
Type of CKD | 2 years
  qualitative variable: pre-dialysis, peritoneal dialysis, hemodialysis
time with CKD | 2 years
  nominal variable: years
time of treatment | 2 years
  nominal variable: years
smoking and alcohol habits | 2 years
  qualitative variable: YES/NO
oral lesions | 2 years
  qualitative variable: uremic odor, xerostomia, taste disorder, petechiae, tongue coating

CONTACTS AND LOCATIONS:
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No